CLINICAL TRIAL: NCT07211386
Title: Efficacy of the Erector Spinae Plane Block for Abdominal Pain From Gastrointestinal Malignancies
Brief Title: The Erector Spinae Plane Block For Gastrointestinal Malignancy Pain Treatment (EGIPT)
Acronym: EGIPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Michael Shalaby, Assistant Professor of Emergency Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 27224
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Malignancy; Pain Control
Keywords: Gastrointestinal malignancy; pain control; nerve block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: 25 patients with gastrointestinal malignancy and abdominal pain who present to any of the four emergency departments within the University of Pennsylvania Health System will be recruited to participate in the study. These patients will have their pain treated with the erector spinae plane block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm -- Erector Spinae Plane Block (Experimental): Patients with gastrointestinal malignancy and abdominal pain will receive the erector spinae plane block for their abdominal pain.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The abdominal viscera, from the stomach to midway through the sigmoid colon, derives its sensory innervation from afferent fibers that travel with, but are distinct from, the sympathetic nerve fibers from the 5th thoracic (T5) to the 2nd lumbar (L2) spinal levels (Moore et al). These fibers converge at the celiac plexus, located near the celiac artery and the aorta. From there, they bifurcate into the paravertebral sympathetic chain and subsequently ascend to the spinal cord and integrate into the central nervous system (Lohse et al). The celiac plexus block is an invasive procedure performed by an interventional anesthesiologist or palliative care specialist to lyse the celiac plexus and has been shown to reduce pain and opiate use in patients suffering from GI malignancy (Ashlock et al). While there are multiple methods to perform a celiac plexus block, it involves a steep needle trajectory either posteriorly through the retroperitoneum or anteriorly through the abdominal wall close

SUMMARY:
This study will target patients with gastrointestinal (GI) malignancy who present to any of 4 Penn Medicine emergency departments (EDs) with intractable abdominal pain. We will offer eligible patients an erector spinae plane block (ESPB), a regional anesthesia technique which is already offered to such patients in the ED at the University of Pennsylvania Healthy System (UPHS), for their intractable abdominal pain. We will compare the outcomes of this prospective cohort of patients to a matched historical control of patients with GI malignancy who were treated in the ED during the same time period as recruitment, but who were not recruited to partake in the study and who were managed with standard of care. Opioid consumption as measured by total milligram morphine equivalents (MMEs) over a 24-hour period and hospital length of stay (LOS) will be compared between cohorts. Additionally, for the ESPB cohort, pain level pre/post ESPB, and functionality and satisfaction with pain management at 24 hours will also be examined.

DETAILED DESCRIPTION:
This study will target patients with gastrointestinal (GI) malignancy who present to any of 4 Penn Medicine emergency departments (EDs) with intractable abdominal pain. We will offer eligible patients an erector spinae plane block (ESPB), a regional anesthesia technique which is already offered to such patients in the ED at the University of Pennsylvania Healthy System (UPHS), for their intractable abdominal pain. We will compare the outcomes of this prospective cohort of patients to a matched historical control of patients with GI malignancy who were treated in the ED during the same time period as recruitment, but who were not recruited to partake in the study and who were managed with standard of care. Opioid consumption as measured by total milligram morphine equivalents (MMEs) over a 24-hour period and hospital length of stay (LOS) will be compared between cohorts. Additionally, for the ESPB cohort, pain level pre/post ESPB, and functionality and satisfaction with pain management at 24 hours will also be examined.

Primary objective: To determine whether patients with GI malignancy receiving an ESPB for intractable abdominal pain consume less opioids (measured in MMEs) in a 24-hour period compared to standard of care analgesia.

Secondary objectives:

To determine whether patients who receive an ESPB have shorter hospital LOS compared to standard of care analgesia.

Within the cohort receiving the ESPB, to determine whether there was a change in pain level as measured by the numeric rating scale (NRS) pre/post block.

Exploratory: Within cohort receiving the ESPB, to determine level of patient satisfaction and functionality as measured by the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R)

Patients with a GI malignancy presenting with intractable abdominal pain. To any of 4 EDs, (1) Hospital of the University of Pennsylvania (HUP), (2) Penn Presbyterian Medical Center (PPMC), (3) Pennsylvania Hospital (PAH), and (4) HUP Cedar (Cedar) Exclusion criteria: pregnant, incarcerated, admissions for serial abdominal examinations, small bowel obstruction, sepsis, altered mental status, hemodynamic instability.

Participants will receive an ESPB, a nerve block performed by injecting anesthetic between a single spinal transverse process and the erector spinae muscle complex (Forero et al). Anesthetic reaches the dorsal nerve root ganglia but also diffuses anteriorly to the paravertebral space which contains the thoracic sympathetic ganglia (Chin et al). Visceral afferent fibers transmit pain signals arising from the stomach to midway through the sigmoid colon utilizing the same anatomical conduit as sympathetic efferent fibers (Moore et al). While physically associated, they travel in the reverse direction of the sympathetic efferents and are functionally distinct. From the abdominal viscera to spinal cord, visceral afferents transmit pain signals first through the peri-aortic autonomic plexuses and prevertebral ganglia, then along the splanchnic nerves to reach the sympathetic trunk, where they travel via the white rami communicantes to reach the spinal nerves of T5 to L2, before finally being conducted centrally. Thus, anesthetizing the thoracolumbar spinal nerves and sympathetic chain, via an ESPB performed between the levels of T5 and L2, should block abdominal visceral pain signaling, and may provide significant analgesia for patients with abdominal pain from GI malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age > 18 years old with GI malignancy presenting to a Penn Medicine ED with intractable abdominal pain.
2. Same-day or recent CT scan of the abdomen / pelvis which demonstrates that the patient's abdominal pain can be reasonably attributed to a malignant source.

Exclusion Criteria:

1. Allergy to ropivacaine or history of local anesthetic systemic toxicity.
2. Pregnancy
3. Incarcerated
4. Patients being admitted for serial abdominal examinations to determine their surgical course.
5. Altered mental status or inability for patient to consent for the procedure
6. Hemodynamic instability
7. Previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | 24 hours
  We will track the amount of opioids consumed within 24 hours by patients who received the erector spinae plane block
Opioid Consumption | 24 hours
  We will track the amount of opioids consumed within 24 hours by participants who receive the erector spinae plane block.

SECONDARY OUTCOMES:
Length of Stay | 1 week
  We will track the total length of stay (emergency department + hospital) for patients who receive the erector spinae plane block
Pain Levels | 30 minutes
  We will track the pain level (measured on a 0-10 Numeric Rating Scale) of participants who receive the erector spinae plane block, and we will compare the difference between their pain immediately before receiving the block and 30 minutes after receiving the block.
Revised American Pain Society Patient Outcome Questionnaire | 24 hours
  We will administer a short 9 question survey graded on a 0-10 scale at 24 hours after participants receive the erector spinae plane block. This survey will assess their pain levels, satisfaction with the erector spinae plane block, ability to move in bed, and ability to move independently out of bed during the 24 hours after they received the erector spinae plane block.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shalaby, MD, Principal Investigator — University of Pennsylvania Department of Emergency Medicine
Locations (4):
- United States (4):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania -- Cedar Avenue, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawel RJ, Kramer JA, Shalaby M. Ultrasound-Guided Erector Spinae Plane Block for Breakthrough Pancreatic and Hepatobiliary Malignancy Pain in the Emergency Department: A Case Series. Clin Pract Cases Emerg Med. 2025 May;9(2):129-133. doi: 10.5811/cpcem.39723. PMID 40402045
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT07211386/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT07211386/ICF_001.pdf